CLINICAL TRIAL: NCT01653704
Title: Learning Crisis Resource Management: Practicing Versus Observational Role in Simulation Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: 20120008-01H
Record Dates: First submitted 2012-07-16; First posted 2012-07-31 (Estimated); Results first posted 2019-01-14 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Focus of Study is Teaching Crisis Resource Management

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- active management of crises scenario (Experimental): participants assigned to actively manage a crisis scenario
  Interventions: Behavioral: active role
- Observer role in crisis scenario (Active Comparator): Observational role in management of crises scenario
  Interventions: Behavioral: observational role

INTERVENTIONS:
Behavioral: observational role — observational role in crisis scenario
  Arms: Observer role in crisis scenario
Behavioral: active role — active role in managing crisis scenario
  Arms: active management of crises scenario

SUMMARY:
The purpose of this study is to compare the effectiveness in learning crisis resource management (CRM) principles when being an active participant in simulation-based education versus being an observer participant. The investigators hypothesize that active participants will improve their CRM skills more than observer participants.

DETAILED DESCRIPTION:
This will be a prospective randomized controlled study. Participants will be randomized to one of two groups with stratification according to their level of training: the active group and the observer group. Each participant of the active group will be paired with one of the participants from the observer group. The active participant will manage individually a simulated crisis scenario (pretest) while the paired observer participant will observe the scenario from outside the simulation room using a video transmission system. Immediately after, both participants will be debriefed by a trained instructor focused on CRM principles. The same active and observer participants will then individually manage another simulated crisis scenario (post-test). Two independent raters, blinded to the study design and to the randomization groups, will review the videos of all scenarios in a random order and rate each participant on their CRM performance using a global rating scale (GRS).

ELIGIBILITY:
Inclusion Criteria:

* emergency medicine residents from the University of Ottawa

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anita Lai, MD, Principal Investigator — University of Ottawa; Sylvain Boet, MD, Principal Investigator — University of Ottawa
Locations (1):
- University of Ottawa Skills and Simulation Centre, Ottawa, Ontario, Canada

REFERENCES:
- [Result] Lai A, Haligua A, Dylan Bould M, Everett T, Gale M, Pigford AA, Boet S. Learning crisis resource management: Practicing versus an observational role in simulation training - a randomized controlled trial. Anaesth Crit Care Pain Med. 2016 Aug;35(4):275-81. doi: 10.1016/j.accpm.2015.10.010. Epub 2016 Mar 14. PMID 26987738

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All emergency medicine residents in postgraduate years 1-5 in both the Royal College of Physicians and Surgeons and College of Family Physician programs at the University of Ottawa were invited to participate in the study.
Period: Overall Study
Arm/Group | Active Management of Crises Scenario | Observer Role in Crisis Scenario
Started | 21 | 21
Completed | 19 | 20
Not Completed | 2 | 1
Not completed — Technical failure during recording | 1 | 1
Not completed — Performance not reflective of training | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Management of Crises Scenario | Observer Role in Crisis Scenario | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Continuous [Mean (Full Range); unit: years] — Population: 2 participants' data experienced technical failure during video recording of performance.
  1 participant's data was excluded from analysis because performance was not reflective of level of training.
  years | NA [NA to NA] — Due to the manner in which data were recorded for this study, baseline data were not associated with the participant study ID, therefore, it is impossible to provide Baseline data per-Arm/Group. | NA [NA to NA] — Due to the manner in which data were recorded for this study, baseline data were not associated with the participant study ID, therefore, it is impossible to provide Baseline data per-Arm/Group. | 29.9 [26 to 43]
Sex/Gender, Customized [Number; unit: participants] — Population: 2 participants' data experienced technical failure during video recording of performance.
  1 participant's data was excluded from analysis because performance was not reflective of level of training.
  participants
    Female | NA — Due to the manner in which data were recorded for this study, baseline data were not associated with the participant study ID, therefore, it is impossible to provide Baseline data per-Arm/Group. | NA — Due to the manner in which data were recorded for this study, baseline data were not associated with the participant study ID, therefore, it is impossible to provide Baseline data per-Arm/Group. | 18
    Male | NA — Due to the manner in which data were recorded for this study, baseline data were not associated with the participant study ID, therefore, it is impossible to provide Baseline data per-Arm/Group. | NA — Due to the manner in which data were recorded for this study, baseline data were not associated with the participant study ID, therefore, it is impossible to provide Baseline data per-Arm/Group. | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Population: 2 participants' data experienced technical failure during video recording of performance.
  1 participant's data was excluded from analysis because performance was not reflective of level of training.
  participants
    Canada | 19 | 20 | 39

OUTCOME MEASURES:

1. Primary Outcome: Total Ottawa GRS Score
Description: The Ottawa GRS scale is a reliable and valid scale used to measure CRM performance in high fidelity simulation. The scale assesses five main CRM categories: leadership, problem solving, situational awareness, resource allocation and communication skills. In addition to these five categories, there is a category on overall performance of the participant. Each category is measured on a 7 point Likert scale with descriptive anchors to provide guidelines on alternating points along the scale. The categorical scores will be summed to give a total score of 6 to 42. Higher values represent a better outcome.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Management of Crises Scenario | Observer Role in Crisis Scenario
Number analyzed (Participants) | 19 | 20
units on a scale | 24.3 (5.4) | 21.8 (4.5)

ADVERSE EVENTS:
Time Frame: Duration the simulation session (1 day)
Arm/Group | Active Management of Crises Scenario | Observer Role in Crisis Scenario
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No